CLINICAL TRIAL: NCT02268981
Title: Effects of an Oxymizer® During Daytime in Patients With Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Dr. med., Schön Klinik Berchtesgadener Land
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12hOXY-ILD2014
Record Dates: First submitted 2014-09-17; First posted 2014-10-20 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Oxymizer; Oxygen conserving device; Conventional nasal cannula (CNC); Idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxymizer® compared to CNC (Experimental): From 7am to 7pm oxygen saturation is measured by a pulse oximeter. One day with conventional nasal cannula, one day with Oxymizer®, one day with Oxymizer® and reduced Oxygen flow (-1l/min). The order of these days is randomized in 6 groups.
  The intervention will be performed on consecutive days and twice during study period.
  Interventions: Device: Oxymizer® compared to CNC

INTERVENTIONS:
Device: Oxymizer® compared to CNC — Oxygen Saturation measurement for 12 h with CNC
  Other Names: Conventional Nasal Cannula (CNC)
Device: Oxymizer® compared to CNC — Oxygen Saturation measurement for 12 h with Oxymizer®
  Other Names: Oxymizer
Device: Oxymizer® compared to CNC — Saturation measurement for 12 h with Oxymizer® by reduced flow rate (-1l/min)
  Other Names: Oxymizer with reduced flow rate (-1l/min)

SUMMARY:
This study will investigate the effects of a reservoir nasal cannula (Oxymizer®) compared to a conventional nasal cannula (CNC) in patients with idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
Patients will be recruited during a 3-week inpatient pulmonary rehabilitation program. They will perform the following three interventions on consecutive days and will repeat them after a week. During these days the time table for prescribed physical activities and therapies will be kept in a comparable fashion.

The following 3 interventions will be performed in randomized order:

Day A: The Patient wears a conventional nasal cannula for 12 h with oxygen flow rate as prescribed during ADL

Day B: The Patient wears the Oxymizer® with prescribed oxygen flow rate for 12 h during ADL

Day C: The patient wears the Oxymizer® with a flow rate reduced by 1l/min in comparison to the prescribed oxygen flow rate, for 12h

The following week the same measurements will be repeated. The mean of the corresponding two measures will be calculated for each approach.

ELIGIBILITY:
Inclusion Criteria:

* IPF patients with indication for long term oxygen therapy ≥ 2l/min
* VC >30% and < 70% pred.

Exclusion Criteria:

* failure to comply with study process
* acute infection

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Difference in oxygen saturation between Oxymizer and conventional nasal cannula | day 1 to 13
  Oxygen Saturation will be measured via pulseoxymetry for 12 hours. On 2 days, mean oxygen Saturation will be reported while using Oxymizer or a conventional nasal cannula, both with similar Oxygen flow. The difference of the mean Oxygen Saturation of 12 hours between both cannulae will be the Primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Dr. med, Study Chair — Schoen Klinik BGL
Locations (1):
- Klinikum Berchtesgadener Land der Schön-Kliniken, Schönau am Königssee, Bavaria, Germany